CLINICAL TRIAL: NCT00393952
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Stratified, Multi-center, 12-Week Study Comparing the Safety and Efficacy of Fluticasone and Formoterol Combination (FlutiForm(tm) 100/10 µg or 250/10 µg Twice Daily) in a Single Inhaler (SkyePharma HFA pMDI) With the Administration of Placebo or Fluticasone (250 µg Twice Daily) and Formoterol (10 µg Twice Daily) Alone in Adolescent and Adult Patients With Moderate to Severe Asthma
Brief Title: New Combination Inhaler (FlutiForm HFA MDI 100/10 µg and 250/10 µg) Versus Fluticasone and Formoterol Administered Alone, and Placebo in Patients With Moderate to Severe Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SkyePharma AG (Industry)
Responsible Party: Skyepharma AG, Skyepharma AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SKY2028-3-004
Record Dates: First submitted 2006-10-27; First posted 2006-10-31 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Asthma
Keywords: Asthma; Fluticasone Propionate; Formoterol Fumarate; Pressurized metered dose inhaler; Hydrofluoroalkane; Moderate-Severe Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (5):
- 1 (Experimental): FlutiForm 250/10
  Interventions: Drug: Fluticasone propionate/Formoterol fumarate 250/10
- 2 (Active Comparator): FlutiForm 100/10
  Interventions: Drug: Fluticasone propionate/Formoterol fumarate 100/10
- 3 (Active Comparator): Fluticasone 250
  Interventions: Drug: Fluticasone propionate 250
- 4 (Active Comparator): Formoterol 10
  Interventions: Drug: Formoterol fumarate 10
- 5 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone propionate/Formoterol fumarate 250/10 — FlutiForm 250/10ug is a HFA pMDI that delivers 125ug of Fluticasone propionate per actuation and 5ug of Formoterol fumarate per actuation. Patients will take 2 actuations BID for 12 weeks.
  Other Names: FlutiForm 250/10
  Arms: 1
Drug: Placebo — Placebo is a HFA pMDI that delivers placebo aerosol. Patients will take 2 actuations BID for 12 weeks.
  Other Names: SKP Placebo
  Arms: 5
Drug: Fluticasone propionate/Formoterol fumarate 100/10 — FlutiForm 100/10ug is a HFA pMDI that delivers 50ug of Fluticasone propionate per actuation and 5ug of Formoterol fumarate per actuation. Patients will take 2 actuations BID for 12 weeks.
  Other Names: FlutiForm 100/10
  Arms: 2
Drug: Fluticasone propionate 250 — Fluticasone 250 is a HFA pMDI that delivers 125ug of Fluticasone propionate per actuation. Patients will take 2 actuations BID for 12 weeks.
  Other Names: Fluticasone 250
  Arms: 3
Drug: Formoterol fumarate 10 — Formoterol 10ug is a HFA pMDI that delivers 5ug of Formoterol fumarate per actuation. Patients will take 2 actuations BID for 12 weeks.
  Other Names: SKP Formoterol 10
  Arms: 4

SUMMARY:
The purpose of this study is to compare the efficacy and safety of the fixed combination asthma drug FlutiForm with its two components administered alone, fluticasone propionate and formoterol fumarate, and with placebo in adult and adolescent patients with moderate to severe asthma.

ELIGIBILITY:
Ages eligible for study: 12 years and above; genders eligible for study: both; prior steroid use: steroid-requiring

Inclusion Criteria:

* History of asthma for at least 12 months.
* Documented use of inhaled corticosteroid for at least 4 weeks prior to Screening Visit Demonstrate FEV-1 of 40-80% of predicted normal values at Screening and Baseline Visit.
* Documented reversibility of 15% within 12 months of Screening visit or at Screening Visit (15% increase from pre-FEV-1 levels following albuterol inhalation or nebulized albuterol administration).
* Symptoms of Asthma during Run-in.
* Females of childbearing potential must have a negative urine pregnancy test at Screening and Baseline Visits. Females are eligible only if they are not pregnant or lactating, and are either sterile or using acceptable methods of contraception
* Must otherwise be healthy.
* Provide written informed consent. Wishes of minors must be respected.

Exclusion Criteria:

* Life-threatening asthma within past year or during Run-In Period.
* History of systemic corticosteroid medication within 3 months before Screening Visit.
* History of omalizumab use within past 6 months.
* History of leukotriene receptor antagonist use, e.g. montelukast, within past week.
* Current evidence or history of any clinically significant disease or abnormality including uncontrolled hypertension, uncontrolled coronary artery disease, congestive heart failure, myocardial infarction, or cardiac dysrhythmia.
* Upper or lower respiratory infection within 4 weeks prior to Screening visit or during Run-In Period
* Significant, non-reversible, pulmonary disease (e.g., chronic obstructive pulmonary disease [COPD], cystic fibrosis, bronchiectasis).
* Known Human Immunodeficiency Virus (HIV)-positive status.
* Smoking history equivalent to "10 pack years".
* Current smoking history within 12 months prior to Screening Visit.
* Current evidence or history of alcohol and/or substance abuse within 12 months prior to Screening visit.
* Patients who are confined in institution.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2006-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Change in Forced Expiratory Volume in 1 s(FEV-1) from Baseline (Week 0) to Week 12. | Week 0 and 12 visits
Discontinuation due to lack of efficacy. | Whole duration of study

SECONDARY OUTCOMES:
Other pulmonary function tests including forced vial capacity (FVC) and peak expiratory flow rate (PEFR). | Whole duration of study
Clinical endpoints (frequency of asthma exacerbations and patient data captured in diary including daily morning and evening PEFR). | Whole duration of study
Serial 12-hour FEV-1 area under the curve (AUC). | Week 0, 2 and 12 visits
Safety variables including adverse events, ECGs clinical laboratory tests and vital signs. | Whole duration of study

CONTACTS AND LOCATIONS:
Locations (60):
- United States (59):
  - Research Center, Pell City, Alabama
  - Research Site, Glendale, Arizona
  - Research Center, Phoenix, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Burbank, California
  - Research Site, Fresno, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Center, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Monterey Park, California
  - Research Site, Palmdale, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Center, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Ormond Beach, Florida
  - Research Center, Panama City, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Tampa, Florida
  - Research Center, Congers, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Round Lake Beach, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Taunton, Massachusetts
  - Research Center, Minneapolis, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Plymouth, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Bozeman, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Brick, New Jersey
  - Research Site, Mount Laurel, New Jersey
  - Research Site, Skillman, New Jersey
  - Research Site, Tinton Falls, New Jersey
  - Research Site, Rockville Centre, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Ashland, Oregon
  - Research Site, Medford, Oregon
  - Research Center, Portland, Oregon
  - Research Center, Upland, Pennsylvania
  - Research Site, Lincoln, Rhode Island
  - Research Center, Anderson, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Center, Fort Worth, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Milwaukee, Wisconsin
- Research Center, Ponce, Puerto Rico